CLINICAL TRIAL: NCT06655298
Title: Ultrasound Guided Erector Spinae Block Versus Quadratus Lumborum Block For Postoperative Pain Relief After Laparoscopic Nephrectomy
Brief Title: Ultrasound Guided Erector Spinae Block Versus Quadratus Lumborum Block For Postoperative Pain ReliefFollowing Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Hamza Sedky, lectuerer, Menoufia University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6/2023ANET44
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pain, Postoperative
Keywords: erector spinae block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups using a closed envelope technique in sequentially numbered opaque envelopes that will be opened before carrying out the block
Who Masked: Participant
Masking Description: closed envelop
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group Q (Experimental): Group Q; (28 patients) Quadratus lumborum block group; patients will receive general anesthesia initially then bilateral QLB type III (anterior subcoastal approach) with a volume of 30 mL of bupivacaine 0.25% for each side taking care that the patient does not receive a local anesthetic dose higher than the maximum allowed (2.5 mg/kg)
  Interventions: Device: US guided block
- group E (Experimental): Group E; (28 patients) Erector spinae plane block; patients will receive general anesthesia initially then bilateral ESPB with a volume of 30 mL of bupivacaine 0.25 % for each side taking care that the patient does not receive a local anesthetic dose higher than the maximum allowed (2.5 mg/kg)
  Interventions: Device: US guided block

INTERVENTIONS:
Device: US guided block — Group Q; (28 patients) Quadratus lumborum block group; patients will receive general anesthesia initially then bilateral QLB type III (anterior subcoastal approach) with a volume of 30 mL of bupivacaine 0.25% for each side taking care that the patient does not receive a local anesthetic dose higher than the maximum allowed (2.5 mg/kg) [9].
  ✓ Group E; (28 patients) Erector spinae plane block; patients will receive general anesthesia initially then bilateral ESPB with a volume of 30 mL of bupivacaine 0.25 % for each side taking care that the patient does not receive a local anesthetic dose higher than the maximum allowed (2.5 mg/kg

SUMMARY:
The aim of this study is to assess the efficacy of Ultrasound guided erector spinae plane block versus quadratus lumborum block for postoperative analgesia in patient undergoing laparoscopic nephrectomy.

DETAILED DESCRIPTION:
The study will be a prospective randomized single-blind study. Patients will be randomized into two groups using a closed envelope technique in sequentially numbered opaque envelopes that will be opened before carrying out the block

The study will be conducted on 56 patients, 28 patients in each group:

Group Q; (28 patients) Quadratus lumborum block group; patients will receive general anesthesia initially then bilateral QLB type III (anterior subcoastal approach) with a volume of 30 mL of bupivacaine 0.25% for each side taking care that the patient does not receive a local anesthetic dose higher than the maximum allowed (2.5 mg/kg) .

✓ Group E; (28 patients) Erector spinae plane block; patients will receive general anesthesia initially then bilateral ESPB with a volume of 30 mL of bupivacaine 0.25 % for each side taking care that the patient does not receive a local anesthetic dose higher than the maximum allowed (2.5 mg/kg)

Data Collection:

Baseline:

1. Patient demographic data
2. Hemodynamics (pulse- heart rate- mean blood pressure), baseline before induction of anesthesia.

Intraoperative:

1. Hemodynamics (pulse- heart rate- mean blood pressure):

   They will be monitored and recorded 5 minutes after induction of anesthesia then every 30 min till end of the surgery.
2. Total analgesic consumption needed to reach target Entropy measurement 40-60%.
3. The anesthetic time (it is the time that starts when the anesthesia provider begins to administer the IV anesthetics and ends with tracheal extubation) and surgical time (starts with skin incision and ends with last suture and putting dressings on).
4. The time taken to perform the block.
5. Number of patients needed ephedrine and/or atropine and total amount of their administration will be recorded.
6. Recovery time (time since anesthetics discontinuation till reaching score 9 of Alderete's criteria).

Postoperative:

1. Time of first call for rescue analgesia.
2. Number of patients requested analgesia postoperative.
3. Visual analogue scale (VAS) on admission to post-anesthetic care unit (PACU), every 30 minutes for next 2 hours, every 2 hours for next 6 hours and every 4 hours for the rest of the 24 hours postoperatively.

   * Discharge from PACU will be according to Postanesthesia Discharge Scoring System[14](Appendix3).
4. Hemodynamics (pulse- heart rate- mean blood pressure)

   They will be assessed as follow:

   • On admission to post-anesthetic care unit (PACU) then every 30 minutes at 30, 60, 90, 120 minutes then every 2 hours for next 6 hours then every 6 hours for remaining 24 hours.
5. Vomiting, nausea and starting time of intestinal movements.
6. Duration of the block (from the injection time of local anesthetic till complete return of sensation).

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II, III scheduled for laparoscopic nepheroctomy

Exclusion Criteria:

* patient refusal bleeding disorders neurological and psychological diseases

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
analgesia | 1 year
  determine the time of first call for rescue analgesia

SECONDARY OUTCOMES:
time | 1 year
  time taken to perform technique

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa mohamed H Sedky, Study Director — lectuerer of anathesia
Locations (1):
- Menoufia University, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No